CLINICAL TRIAL: NCT01489670
Title: Observational Study of Lumigan® 0.01% Treatment for Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/032
Record Dates: First submitted 2011-12-01; First posted 2011-12-12 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumigan® 0.01%: Patients with primary open-angle glaucoma or ocular hypertension treated with Lumigan® 0.01% in clinical practice.
  Interventions: Drug: bimatoprost 0.01% ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost 0.01% ophthalmic solution — Patients with primary open-angle glaucoma or ocular hypertension treated with Lumigan® 0.01% in clinical practice.
  Other Names: Lumigan® 0.01%

SUMMARY:
This study will assess the efficacy, safety, tolerability and persistence of use of Lumigan ® 0.01% in patients diagnosed with primary open-angle glaucoma or ocular hypertension who are treated per routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma or ocular hypertension
* Lumigan® 0.01% prescribed either as monotherapy or adjunctive to beta-blocker therapy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary open-angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Bülach, Canton of Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with primary open-angle glaucoma or ocular hypertension treated with Lumigan® 0.01% in clinical practice. There was no investigational drug administered in this study.
Period: Overall Study
Arm/Group | Lumigan® 0.01%
Started | 387
Completed | 334
Not Completed | 53

BASELINE CHARACTERISTICS:
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 387
Age, Customized [Number; unit: Participants]
  18 to 30 Years | 1
  31 to 40 Years | 3
  41 to 50 Years | 28
  51 to 60 Years | 53
  61 to 70 Years | 113
  71 to 80 Years | 120
  81 to 90 Years | 62
  >=91 Years | 5
  Missing data | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237
  Male | 150

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Baseline
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left and right eye at Baseline.
Time Frame: Baseline
Population: All participants with complete data available for IOP.
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 335
mm Hg
  Right Eye (n=334) | 22.0 [10.0 to 50.0]
  Left Eye | 22.0 [7.0 to 52.0]

2. Secondary Outcome: Physician Evaluation of Efficacy Using a 5-Point Scale
Description: The physician evaluated efficacy using a 5-point scale (IOP lower than the target, Target IOP reached, IOP decreased but target not reached, IOP increased or No change). The number of participants in each category is reported.
Time Frame: Week 12
Population: All participants with data available for this outcome measure.
Measure: Number; unit: Participants
Units Other Than Participants: Eyes
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 341
Number analyzed (Eyes) | 405
Participants
  IOP lower than target | 87
  Target IOP reached | 187
  IOP decreased but target not reached | 64
  IOP increased | 6
  No Change | 15

3. Secondary Outcome: Patient Evaluation of Tolerability of Treatment Using a 4-Point Scale
Description: Patients evaluated their tolerability of treatment using a 4-point scale (very good, good, moderate, and poor). The number of participants in each category is reported.
Time Frame: Week 12
Population: All participants with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 324
Participants
  Very good | 157
  Good | 144
  Moderate | 7
  Poor | 16

4. Secondary Outcome: Physician Evaluation of Tolerability of Treatment
Description: The physician evaluated the patient's tolerability of treatment using a 4-point scale (very good, good, moderate, and poor). The percentage of participants assessed in each category is reported.
Time Frame: Week 12
Population: All participants with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 333
Participants
  Very good | 174
  Good | 141
  Moderate | 12
  Poor | 6

5. Secondary Outcome: Physician Reported Reasons for Early Discontinuation of Treatment
Description: The number of patients who discontinued from treatment by category is reported. More than one reason may apply to each patient.
Time Frame: 12 Weeks
Population: All participants who discontinued treatment early.
Measure: Number; unit: Participants
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 53
Participants
  Unacceptable ocular tolerability | 28
  Patient decision to withdraw from study | 21
  Insufficient IOP control | 18
  Physician decision to withdraw patient from study | 8
  Patient lost to follow up | 1
  Other reason | 6
  Missing data | 1

6. Secondary Outcome: Number of Patients Continuing Treatment After 12 Weeks
Description: The number of patients continuing treatment after 12 weeks was determined by the physician answering yes to the question: Is the patient continuing on Lumigan® 0.01% treatment?
Time Frame: Week 12
Population: All participants with data available for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 345
Participants | 302

7. Primary Outcome: Intraocular Pressure (IOP) at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left and right eye at the Final Visit at approximately Week 12. The lower the IOP values the greater the improvement.
Time Frame: Week 12
Population: All participants with complete data available for IOP.
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Lumigan® 0.01%
Number analyzed (Participants) | 335
mm Hg
  Right Eye (n=334) | 16.0 [1.0 to 32.0]
  Left Eye | 16.0 [8.0 to 28.0]

ADVERSE EVENTS:
Arm/Group | Lumigan® 0.01%
Serious Adverse Events (participants affected / at risk) | 0/387
Other Adverse Events (participants affected / at risk) | 148/387
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumigan® 0.01% (N=387)
Conjunctival hyperaemia (Eye disorders) | 75
Eye irritation (Eye disorders) | 46
Eye pruritus (Eye disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.